CLINICAL TRIAL: NCT01760369
Title: Observation Study of the: Effect of Head Rotation in Prone Position on Regional Cerebral Oxygen Saturation (rSO2) in Anesthetized Patients.
Brief Title: Study of the: Effect of Head Rotation in Prone Position on Regional Cerebral Oxygen Saturation.
Acronym: NIRS
Status: Completed | Type: Observational
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Johnny Andersen, Medical Doctor, Glostrup University Hospital, Copenhagen
Other Study IDs: NIRS-JDHA-12
Record Dates: First submitted 2012-12-20; First posted 2013-01-04 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-01

CONDITIONS: Regional Cerebral Oxygen Saturation During Head Rotation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether head rotation in prone positon affects regional cerebral oxygenation (rSO2)in anesthetized patients undergoing lower back surgery.

ELIGIBILITY:
Inclusion Criteria:

* Lower back surgery
* Age [18-80]
* ASA group I-III
* free and painless movement of the neck (including flexion, extension and rotation)

Exclusion Criteria:

* Pain during neck movement as mentioned under inclusion criteria.
* known history of cervical spine pathology or pathology of central nervous system including cerebrovascular disease
* any stenosis of the carotid vessels or known symptoms associated with such
* BMI > 35

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing lowerback surgery under universal anesthesia at Glostrup Hospital, Copenhagen.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in regional cerebral oxygenation (rSO2) | 1 day
  Before, during and immediately after awaking from anesthesia

SECONDARY OUTCOMES:
Post anesthetic complications | 1 day
  During stay at the post anesthetic care unit. Any new neurological symptoms, pain from the neck, visual symptoms etc.

CONTACTS AND LOCATIONS:
Overall Officials: Johnny DH Andersen, Doctor, Principal Investigator — Doctor
Locations (1):
- Glostrup Hospital, Copenhagen, Glostrup kommune, Denmark

REFERENCES:
- [Derived] Andersen JD, Baake G, Wiis JT, Olsen KS. Effect of head rotation during surgery in the prone position on regional cerebral oxygen saturation: A prospective controlled study. Eur J Anaesthesiol. 2014 Feb;31(2):98-103. doi: 10.1097/EJA.0000000000000028. PMID 24335413